CLINICAL TRIAL: NCT00703274
Title: Preventing Recurrence of Thromboembolic Events Through Coordinated Treatment in the District of Columbia
Acronym: PROTECT DC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Chelsea Kidwell, M.D., Medical Director, Georgetown University Stroke Center, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: U54NS057405 (NIH); 1U54NS057405-01A1 (NIH)
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Stroke
Keywords: ischemic stroke; stroke; cerebrovascular stroke; cerebrovascular accident; CVA; community health services; community health workers; navigators; health education; barriers to care; healthcare access; healthcare disparities
MeSH Terms: conditions — Stroke; Ischemic Stroke; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navigation Group (Experimental): Participants enrolled in this group will receive education concerning primary and secondary PROTECT DC goals. Primary PROTECT DC goals adhere to the following medication directives: 1) Anti-hypertensive, 2) Lipid Lowering, 3) Anti-Coagulant, and 4) Anti-Diabetic. PROTECT DC secondary goals include the following behaviors 1) Smoking Cessation, 2) Consuming an AHA Diet, 3) Regular Exercise, and 4) Knowledge of Stroke Risk and Warning Signs. Participants will also receive assistance with overcoming resource-related barriers to the PROTECT DC goals.
  Interventions: Behavioral: PROTECT DC
- Control Group (No Intervention): Participants enrolled in this group will receive periodic follow up through mailings, phone calls etc to ensure availability for 1 year assessment.

INTERVENTIONS:
Behavioral: PROTECT DC — PROTECT DC facilitates the initiation of secondary prevention behaviors in an attempt to prevent the recurrence of stroke among participants. The program trains a lay person, called a stroke navigator, to provide participants with education on secondary prevention behavior and to navigate the health and human service system, which will assist participants in obtaining the necessary services and programs to engage in secondary prevention behaviors.
  Other Names: navigator model; navigation intervention; community health worker intervention
  Arms: Navigation Group

SUMMARY:
The purpose of this study is to refine and evaluate the Preventing Recurrence of Thromboembolic Events through Coordinated Treatment in the District of Columbia (PROTECT DC) intervention. PROTECT DC is a program consisting of in-hospital education coupled with community-based "stroke navigators" and is designed to reduce the rate of vascular events or death in a population of underserved individuals with stroke.

DETAILED DESCRIPTION:
Despite significant advances in the prevention and treatment of cerebrovascular disease in the last few decades, stroke remains the third leading cause of death and the leading cause of adult disability in the United States. For the population that has experienced a cerebrovascular event, the risk of future stroke is greatly increased. The initiation of effective secondary prevention strategies is most effective when implemented early (before disabling stroke occurs), monitored frequently, and maintained long-term after a cerebrovascular event.

The Preventing Recurrence of Thromboembolic Events through Coordinated Treatment in the District of Columbia (PROTECT DC) intervention uses stroke navigators to help people who have suffered a stroke implement secondary prevention strategies. Stroke navigators are lay persons trained to provide education on secondary prevention behavior, and trained to navigate the health and human service system. The goals are to help individuals who have had a stroke obtain the necessary services and programs to engage in secondary prevention behaviors and, ultimately, to prevent the recurrence of stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized due to ischemic stroke* or intercurrent ischemic stroke* event within the past 30 days OR Transient ischemic attack, confirmed by stroke neurologist.
* Atherogenic etiology(large vessel, small vessel, cryptogenic with at least one stroke risk factor, or embolic stroke due to atherogenic cardiac disease) as defined by TOAST criteria.
* Community dwelling prior to stroke
* Resides within the District of Columbia or closely nearby (preferably within 10 miles of the DC border)
* Expected to reside within the District of Columbia or closely nearby (preferably within 10 miles of DC border)
* Caregiver or interested party available, if moderately or severely disabled (not required to actually reside with participant)
* Sufficient number of collateral contacts to assure follow-up. Defined as: Preferred: at least 6 contacts; and No fewer than 3 contacts (unless approved by study PI/co-PI/co-I)
* Judged likely to return to community setting at completion of post-acute care.

Exclusion Criteria:

* Non-atherogenic cause of stroke
* NIHSS > 20
* Any medical condition that would limit participation in follow up assessments
* Baseline dementia per informant report (AD8) or screening assessment (Short Blessed Memory Orientation Concentration Test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2008-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Low Density Lipoprotein Value | 1 year
Systolic Blood Pressure Value | 1 year
Hemoglobin A1C Value | 1 year
Pill count of antiplatelet therapy medications | 1 year

SECONDARY OUTCOMES:
Smoking Cessation Status | 1 year
AHA Diet Status | 1 year
Exercise Status | 1 year
Stroke Knowledge Level | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Dromerick, MD, Principal Investigator — National Rehabilitation Hospital, Georgetown University; Chelsea S. Kidwell, MD, Principal Investigator — Washington Hospital Center, National Rehabilitation Hospital, Georgetown University
Locations (6):
- United States (6):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - National Rehabilitation Hospital, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Providence Hospital, Washington D.C., District of Columbia
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia

REFERENCES:
- [Background] Dromerick AW, Gibbons MC, Edwards DF, Farr DE, Giannetti ML, Sanchez B, Shara NM, Fokar A, Jayam-Trouth A, Ovbiagele B, Kidwell CS. Preventing recurrence of thromboembolic events through coordinated treatment in the District of Columbia. Int J Stroke. 2011 Oct;6(5):454-60. doi: 10.1111/j.1747-4949.2011.00654.x. PMID 21951411